CLINICAL TRIAL: NCT06952036
Title: The Epidemic Status and Development Trend of Hepatitis C Virus Infection in Pregnant Women in Xi'an: A 10-Year Retrospective Study
Brief Title: The Epidemic Status and Development Trend of Hepatitis C Virus Infection in Pregnant Women in Xi'an
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, He Yingli, Director of Department of Infectious Diseases, the First Affiliated Hospital of Jiaotong University, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: XJTU1AF2024LSYY-413
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: HCV Infection; HCV Elimination
Keywords: Hepatitis C; HCV elimination; Women of childbearing age
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women who had an antenatal visit or gave birth between 2014 and 2023.
  Interventions: Procedure: Standard Direct-acting antivirals (DAA) treatment procedures for patients with hepatitis C

INTERVENTIONS:
Procedure: Standard Direct-acting antivirals (DAA) treatment procedures for patients with hepatitis C — Initiated Standard DAA treatment among HCV RNA positive patients.

SUMMARY:
The objectives of this study are to improve HCV linkage-to-care in Chinese women and provide theoretical basis for the scientific formulation of HCV prevention and control strategies for pregnant women.

To understand the epidemiological changes and status of hepatitis C virus (HCV) infection in pregnant women in Shaanxi province in recent 10 years, and to analyze the main influencing factors of hepatitis C infection in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women or parturient women confirmed by blood HCG test.
2. Patients aged 18 years old and above.
3. Patients with HCV antibody seropositive or HCV RNA positive from 2014-2023.

Exclusion Criteria:

1. Patients without valid telephone numbers.
2. Duplicate records: For duplicate records of the same pregnant woman, only one record should be kept.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women who had an antenatal visit or gave birth between 2014 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relink rate | From enrollment to the end of treatment at 12 weeks
  The percentage of patients receiving DAA treatment among the diagnosed but untreated patients.